CLINICAL TRIAL: NCT05947422
Title: CT Quantitative Assessment of Interstitial Lung Disease Using Visual Score and Lung Densitometry Methods and Its Correlation With Pulmonary Function Tests
Brief Title: CT Quantitative Assessment of Interstitial Lung Disease
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ramy Mohammed Ahmed, lecturer and consultant of diagnostic an dintervention radiology, Assiut University
Other Study IDs: ILD-CT
Record Dates: First submitted 2023-06-13; First posted 2023-07-17 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Spirometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: High resolution CT Chest — CT chest in our institution will be done with standard high resolution protocol . No I.V contrast will be given. Scans will be obtained during full inspiration in supine position from the thoracic inlet to the level of the diaphragm.
  Patients with CT chest performed outside our institution will be reviewed in DICOM format and assessed for its compatibility to be integrated into the computer-based analysis software.
Diagnostic Test: Spirometry — Spirometry will be performed using standard techniques according to ATS-ERS criteria 2019 . Spirometry device (Zan 300, NSPIRE HEALTH GMBH Co.) will be used. Percentage predicted values (%pred) will be calculated based on reference values for healthy adults. All patients will be required to undergo spirometry in a reproducible way, and the best values will be reported. Spirometry should meet international acceptability and repeatability standards

SUMMARY:
Interstitial lung disease (ILD) refers to a broad category of heterogeneous lung diseases with different etiologies and features characterized by inflammation and fibrosis of the lung parenchyma and manifested as exertional dyspnea, interstitial patterns on high resolution computed tomography (HRCT), and abnormal pulmonary function tests (PFTs) The aim of this study is to investigate is there any correlation between changes seen in the lung parenchyma by HRCT and the pulmonary functions of the patients.

DETAILED DESCRIPTION:
This study will utilize a cross-sectional prospective study design in a single institution to investigate the correlation between CT chest findings including lung densitometry and pulmonary function test results in patients with ILD.

The study population will consist of consecutive patients diagnosed with ILD recruited from the pulmonary clinic or inpatient service.

High resolution CT chest and pulmonary function tests are routine diagnostic tests used for diagnosis of interstitial lung disease .

both tests are non invasive for the patient and will be acquired for all patients and then their results will be correlated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ILD (based on clinical, radiological, and pulmonary function criteria +/- histopathological criteria).
* Availability of CT chest DICOM images and pulmonary function test results (within a 2-weeks period from each other).

Exclusion Criteria:

* Pregnancy
* Pulmonary edema.
* Primary pulmonary hypertension;
* Chronic obstructive pulmonary disease
* Congestive heart failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of consecutive patients diagnosed with ILD recruited from the pulmonary clinic or inpatient service. The diagnosis of ILD will be based on American Thoracic Society/European Respiratory Society (ATS/ERS) classification system for ILD.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
CT visual Warrick score (measured by points) | baseline
  Warrick score is calculated as follow : A point value will be given to each abnormality i.e ground-glass appearance (areas of hazy opacity in the lung that do not obscure the underlying bronchial structures) = 1, irregular pleural margins = 2, septal/subpleural lines = 3, honeycombing (usually 3-10 mm in diameter and have thick walls) = 4, and subpleural cysts = 5. In each patient, the "severity of disease" score will be obtained by adding single point values (maximal severity score 15).
  An "extent of disease" score is obtained by counting the number of bronchopulmonary segments involved for each abnormality as follows ; one to three segments scored as 1, four to nine segments scored as 2, and more than nine segments scored as 3 (maximal extent score 15).
  The severity and extent of disease will be then calculated as the total Warrick score (range from 0 to 30)
Total lung volume, Volume of lung occupied by low attenuation areas, Volume of lung occupied by high attenuation areas, Volume of normal lung areas and volume of consolidation areas | baseline
  Total lung volume , volume of the lung occupied by low attenuation areas (attenuation values from -1024 to -950 HU; representing emphysema), volume of normally attenuated lung (from -949 to -700 HU; corresponds to healthy lung tissue) and volume of the lung occupied by high attenuation areas (between - 699 and - 250 HU) ; it represents the lung parts which are more dense than healthy lung); volume of lung with density from -249 to +40 HU, this group corresponds to areas with further increase in density, including the semi-consolidation and consolidation.
Percentage of the lung occupied by low attenuation areas, percentage of normal lung, percentage of the lung occupied by high attenuation areas and percentage of consolidation areas. | baseline
  Percentage of the lung occupied by low attenuation areas (attenuation values from -1024 to -950 HU), percentage of normal lung (from -949 to -700 HU), percentage of the lung occupied by high attenuation areas (between - 699 and - 250 HU) and percentage of consolidation areas (from -249 to +40 HU) in each lung and in each lobe.
Mean lung density of each lung, both lungs and every lobe in Hounsfield unit (HU) | baseline
  Mean lung density of each lung , both lungs and each lung lobe (e.g., upper, middle, and lower lobes) will be measured in Hounsfield unit (HU).
Forced vital capacity (FVC) | baseline
  Forced vital capacity (FVC) will be measures using spirometer and expressed as percentage.
Forced expiratory volume in 1 second (FEV1) | baseline
  Forced expiratory volume in 1 second (FEV1)
FEV1/FVC ratio | baseline
  FEV1/FVC ratio will be measures
O2 saturation | baseline
  O2 saturation is measured in percentage (SpO2) using pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Ramy M Ahmed, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Asyut Governorate, Egypt